CLINICAL TRIAL: NCT01010841
Title: Multi-center, Randomized Intervention to Compare the Effects of 2 Dietary Programs on Cardiometabolic Risk Factors in Subjects With Metabolic Syndrome
Brief Title: Trial of Two Dietary Programs on Cardiometabolic Risk Factors in Subjects With Metabolic Syndrome
Acronym: HMS4
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaProteomics LLC (Industry)
Collaborators: University of Florida (Other); University of Connecticut (Other); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMS4-MUL-CT
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Metabolic Syndrome; Overweight; Obesity; Hypercholesterolemia
Keywords: Metabolic syndrome; Serum lipid; Dietary intervention; Lifestyle modification; Glycemic load; Phytochemical; Hops; Acacia; Mediterranean diet; Kinase modulator
MeSH Terms: conditions — Metabolic Syndrome; Overweight; Obesity; Hypercholesterolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-glycemic-load diet (Active Comparator): Modified Mediterranean-style low-glycemic-load diet
  Interventions: Other: Low-glycemic-load diet
- Low-glycemic-load diet + medical food (Experimental): Modified Mediterranean-style, low-glycemic-load diet + medical food
  Interventions: Dietary Supplement: UltraMealPlus 360 (Medical food); Other: Low-glycemic-load diet

INTERVENTIONS:
Dietary Supplement: UltraMealPlus 360 (Medical food) — Specific phytochemicals (soy protein, phytosterols, rho iso-alpha acids and proanthocyanidins; PED)
  Other Names: UltraMealPlus 360
  Arms: Low-glycemic-load diet + medical food
Other: Low-glycemic-load diet — Modified Mediterranean-style low-glycemic-load diet

SUMMARY:
The objective of this study was to investigate from 3 sites (University of Connecticut, University of Florida, and University of California, Irvine) whether enhancement of a modified Mediterranean-style, low glycemic load diet (MED) with specific phytochemicals (soy protein, phytosterols, rho iso-alpha acids and proanthocyanidins; PED) could improve cardiometabolic risk factors in women with metabolic syndrome.

DETAILED DESCRIPTION:
As the worldwide dietary pattern becomes more westernized, the metabolic syndrome is reaching epidemic proportions. Lifestyle modifications including diet and exercise are recommended as first-line intervention for treating metabolic syndrome. Previously, we reported that specific phytochemical supplementation for 12 weeks (soy protein, phytosterols, rho iso-alpha acids and proanthocyanidins) increased the effectiveness of the modified Mediterranean-style low glycemic load dietary program on variables associated with metabolic syndrome and CVD in subjects with metabolic syndrome and elevated LDL cholesterol. In this study, we propose to conduct a multi-center randomized trial to confirm our previous findings.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25 and <45
* LDL >100 mg/dl
* TG ≥150 and <400 mg/dl
* meet 2 or more of the following 4 criteria:

  * HDL <50 mg/dl
  * blood pressure ≥130/85 mmHg (or diagnosed hypertension on medication)
  * fasting glucose ≥100 mg/dl and <150 mg/dl
  * waist circumference >35 inches

Exclusion Criteria:

* Medical History and Concurrent Diseases

  1. Over the preceding 4 weeks, initiation or cessation of regular exercise
  2. Over the preceding 4 weeks, involvement in a significant diet or weight loss program such as Atkin's diet program, a very low calorie liquid program (such as Optifast, Medifast, and HMR), or any diet that has led to a weight loss of 10% of body weight over a period of 6 weeks
  3. Use of blood sugar lowering medications including thiazolidinedione class of oral medications including Avandia (rosiglitazone), Avandamet (metformin/rosiglitazone), Actos (pioglitazone), metformin (Glucophage, Fortamet, Riomet) or insulin over the preceding 12 weeks
  4. Over the preceding 4 weeks, regular use of Kaprex® or Kaprex AI® at least 3 days/week
  5. Over the preceding 4 weeks, regular use of NSAIDs (i.e. ibuprofen, celecoxib, etc.) at least 3 days per week
  6. Over the preceding 12 weeks, use of cholesterol lowering medications, either by prescription (statins, etc.) or over-the-counter (gugulipids, niacin, etc.)
  7. Over the preceding 12 weeks, use of oral or injectable corticosteroids, such as prednisone
  8. Current use of oral anticoagulants such as Coumadin or injectable anticoagulants such as Heparin or Low Molecular Weight Heparin
  9. Use of electronic implants such as pacemakers, defibrillators, nerve stimulators
  10. Allergy to one or more of the ingredients in the investigational products
  11. Poorly controlled hypertension (blood pressure above 155/95)
  12. History of significant liver or kidney disease (recent or ongoing hepatitis, cirrhosis, glomerulonephritis, dialysis treatment, etc.)
  13. History of serious heart disease (heart attack, angina, cardiac surgery, arrhythmia, or congestive heart failure)
  14. History of deep vein thrombosis or pulmonary embolus (blood clot to lungs)
  15. History of autoimmune diseases such as inflammatory bowel disease (Crohn's disease, and/or ulcerative colitis), multiple sclerosis, rheumatoid arthritis, systemic lupus erythematosus, polymyositis, scleroderma and thyroiditis
  16. History of eating disorder (anorexia nervosa or bulimia) in preceding 5 years
  17. History of alcoholism or drug addiction in the preceding 5 years
  18. History of serious mental illness
  19. History of attempted suicide in past 10 years
  20. Untreated endocrine, neurological, or infectious disorder
  21. Diagnosis of Human Immunodeficiency Virus (HIV) or Acquired HIV (AIDS)
  22. Current cancer or a history of cancer (except skin cancer)
  23. Pregnancy or lactation
  24. If female of childbearing potential, unwillingness to practice a reliable method of birth control (i.e. physical sperm barriers or hormonal therapies)
  25. Any other sound medical, psychiatric and/or social reason as determined by the Principal Investigator (PI).
* Physical and Laboratory Test Findings

  1. TG ≥ 400 mg/dl
  2. abnormal blood count (Hct < 30 or > 47%, WBC < 3,000 or > 12,000, platelets <140 or > 500)
  3. abnormal kidney function test(s) (BUN > 30 mg/dL or creatinine > 1.5 mg/dL) or liver function test(s) (bilirubin total > 2.0 mg/dL, ALT > 75 IU/L, AST > 75 IU/L; Alk Phos > 130 IU)
  4. fasting glucose >150 mg/dL, serum calcium (>10.5 mg/dL), positive pregnancy test (ß-hCG in blood)

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
TG-to-HDL ratio | Baseline, 8 weeks, 12 weeks

SECONDARY OUTCOMES:
Components of metabolic syndrome (TG, HDL, resolution of MetS) | Baseline, 8 weeks, 12 weeks
Glucose intolerance (fasting glucose/insulin, leptin, HbA1c, HOMA score) | Baseline, 8 weeks, 12 weeks
CVD risk factors (cholesterol, LDL, chol/HDL, apoAI, apoB, apoAII, apoCII, apoCIII, apoE, homocysteine, RBC fatty acids, Framingham risk score) | Baseline, 8 weeks, 12 weeks
Inflammatory cytokines (TNF-alpha, IL-6, sICAM, sVCAM, MCP1) | Baseline, 8 weeks, 12 weeks
Body composition (weight, BMI, % body fat, % lean mass, waist-to-hip ratio, DEXA scanning) | Baseline, 8 weeks, 12 weeks
Subjective assessment (MOS-MCS/PCS questionnaires, VAS-satiety/craving questionnaires) | baseline, then every 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Lerman, MD/PhD, Study Director — MetaProteomics LLC; Mark McIntosh, MD, Principal Investigator — University of Florida; Maria Luz Fernandez, PhD, Principal Investigator — University of Connecticut; Wadie Najm, PhD, Principal Investigator — University of California at Irvine
Locations (1):
- Mark McIntosh MD, Jacksonville, Florida, United States

REFERENCES:
- [Result] Jones JL, Fernandez ML, McIntosh MS, Najm W, Calle MC, Kalynych C, Vukich C, Barona J, Ackermann D, Kim JE, Kumar V, Lott M, Volek JS, Lerman RH. A Mediterranean-style low-glycemic-load diet improves variables of metabolic syndrome in women, and addition of a phytochemical-rich medical food enhances benefits on lipoprotein metabolism. J Clin Lipidol. 2011 May-Jun;5(3):188-196. doi: 10.1016/j.jacl.2011.03.002. Epub 2011 Mar 11. PMID 21600524
- [Result] Fernandez ML, Jones JJ, Ackerman D, Barona J, Calle M, Comperatore MV, Kim JE, Andersen C, Leite JO, Volek JS, McIntosh M, Kalynych C, Najm W, Lerman RH. Low HDL cholesterol is associated with increased atherogenic lipoproteins and insulin resistance in women classified with metabolic syndrome. Nutr Res Pract. 2010 Dec;4(6):492-8. doi: 10.4162/nrp.2010.4.6.492. Epub 2010 Dec 28. PMID 21286407
- [Result] Ackermann D, Jones J, Barona J, Calle MC, Kim JE, LaPia B, Volek JS, McIntosh M, Kalynych C, Najm W, Lerman RH, Fernandez ML. Waist circumference is positively correlated with markers of inflammation and negatively with adiponectin in women with metabolic syndrome. Nutr Res. 2011 Mar;31(3):197-204. doi: 10.1016/j.nutres.2011.02.004. PMID 21481713
- [Result] Barona J, Jones JJ, Kopec RE, Comperatore M, Andersen C, Schwartz SJ, Lerman RH, Fernandez ML. A Mediterranean-style low-glycemic-load diet increases plasma carotenoids and decreases LDL oxidation in women with metabolic syndrome. J Nutr Biochem. 2012 Jun;23(6):609-15. doi: 10.1016/j.jnutbio.2011.02.016. Epub 2011 Jul 19. PMID 21775117
- [Result] Jones JL, Comperatore M, Barona J, Calle MC, Andersen C, McIntosh M, Najm W, Lerman RH, Fernandez ML. A Mediterranean-style, low-glycemic-load diet decreases atherogenic lipoproteins and reduces lipoprotein (a) and oxidized low-density lipoprotein in women with metabolic syndrome. Metabolism. 2012 Mar;61(3):366-72. doi: 10.1016/j.metabol.2011.07.013. Epub 2011 Sep 23. PMID 21944261
- [Result] Jones JL, Park Y, Lee J, Lerman RH, Fernandez ML. A Mediterranean-style, low-glycemic-load diet reduces the expression of 3-hydroxy-3-methylglutaryl-coenzyme A reductase in mononuclear cells and plasma insulin in women with metabolic syndrome. Nutr Res. 2011 Sep;31(9):659-64. doi: 10.1016/j.nutres.2011.08.011. PMID 22024489
- [Result] Jones JL, Ackermann D, Barona J, Calle M, Andersen C, Kim JE, Volek JS, McIntosh M, Najm W, Lerman RH, Fernandez ML. A Mediterranean low-glycemic-load diet alone or in combination with a medical food improves insulin sensitivity and reduces inflammation in women with metabolic syndrome. British Journal of Medicine & Medical Research 1(4):356-370, 2011.